CLINICAL TRIAL: NCT05055973
Title: Optical Coherence Tomography Angiography Insights in Choroidal Neovascular Membrane, Morphological Characteristics and Correlation With Structural Optical Coherence Tomography.
Brief Title: OCTA Insights in CNVM, Morphological Characteristics and Correlation With Structural OCT.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Mahmoud A. Abdallah, Principle Investigator, Assiut University
Other Study IDs: OCTAIICNMMCACWSOCT
Record Dates: First submitted 2021-09-12; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To suggest a novel classification of choroidal neovascular membrane based on optical coherence tomography angiography and to correlate morphological characteristics based on optical coherence tomography with clinical criteria of disease activity.

DETAILED DESCRIPTION:
Choroidal neovascularization is an important path biologic mechanism encountered in a variety of chorio-retinal diseases. Choroidal neo-vascularization represents new blood vessel growth from the choroid that extends into the sub-retinal pigment epithelium, or sub-retinal space, or a combination of both. There is some evidence that the clinical findings and angiographic appearance of choroidal neo-vascular membrane correlate with the growth pattern. Choroidal neo- vascularization dynamic evolution includes initiation, inflammatory active, and inflammatory inactive stages.

It can be assumed that there is a risk of choroidal neo-vascular membrane development in any case where the integrity of Bruch's membrane or the retinal pigment epithelium is impaired. The most common cause of choroidal neo-vascular membrane is indisputably age-related macular degeneration, but choroidal neo-vascular membrane may also occur secondary to many other etiologies, such as pathological myopia, angioid streaks, uveitis, infection, and traumatic Bruch's membrane-retinal pigment epithelium defects, and idiopathic cases where no etiology can be detected.

Growth pattern:

Although no two choroidal neo-vascular membrane growth patterns are exactly alike, choroidal neo-vascular membrane grows in the plane between the retinal pigment epithelium and the Bruch membrane, between the retina and retinal pigment epithelium, or a combination of both (combined pattern). There is a retinal vascular contribution in approximately 6% of choroidal neo-vascular membrane . The new blood vessels are capillary-like and, with time, become arterial and venular.

Imaging modalities:

Fundus fluorescein angiography with dye injection is considered the gold standard for detecting choroidal neo-vascular membrane and assessing its activity. However, Fundus fluorescein angiography is time consuming and invasive, resulting in varying degrees of patient discomfort, including anaphylactic reactions that can occur during and/or after fundus fluorescein angiography. A total of 4.8% patients were reported to have experienced adverse events after the fundus fluorescein angiography, including nausea (2.9%), vomiting (1.2%), and flushing/itching (0.5%).

Optical coherence tomography has become an important non-invasive and quick method to diagnose and monitor disease activity during anti- vascular endothelial growth factor treatment by revealing the fate of active choroidal neo-vascular membrane such as intra- and sub-retinal fluid accumulation and retinal thickening. On optical coherence tomography CNV appears as sub-retinal or sub-retinal pigment epithelium hyper reflective material with limited differentiation between unreactive fibrous and/or active neo-vascular tissue. Retreatment decisions are mainly based on assessment of extravascular fluid and not on an analysis of neo-vascular activity.

Optical coherence tomography angiography offers a breakthrough in diagnostic imaging by allowing non-invasive visualization of retinal and choroidal vascular flow via motion-contrast imaging. Optical coherence tomography angiography provides depth-resolved visualization of the retinal and choroidal vasculature without the need for dye injection. The technology has been applied for the diagnosis and monitoring of choroidal neo-vascular membrane in age-related macular degeneration. Optical coherence tomography angiography has described features of myopic choroidal neo-vascular membrane and demonstrated its high sensitivity and specificity for neo-vascular detection. Optical coherence tomography angiography is a new noninvasive imaging modality, based on high-frequency scanning for the detection of blood cell movement. This imaging modality takes advantage of the optical coherence tomography capacity to generate images by measuring the amplitude and delay of reflected and backscattered light. Multiple repeated scans are carried out in the same retinal location, and the images obtained are compared to identify the signal differences between two consecutive scans. Because the retina is a static structure, it is reasonable to suppose that these changes are imputable to the blood flow. This precise and non-invasive imaging modality offers novel diagnostic opportunities to fill the current gap between invasive vascular and non- invasive structural imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with all types of CNV, previously treated or naïve.

Exclusion Criteria:

* The presence of prominent media opacity.
* Significant cataract.
* Poor fixation.
* Any other factor that interferes with obtaining good-quality OCT/OCTA images.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with choroidal neovascular membrane, naive or previously treated.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Morphological characters of choroidal neovascular membrane | One year
  To describe morphological criteria of choroidal neovascular membrane using optical coherence tomography angiography (OCTA).

SECONDARY OUTCOMES:
Correlation between morphological characters of choroidal neovascular membrane and disease activity | One year
  To correlate the morphological characters of choroidal neovascular membrane and clinical criteria of disease activity

CONTACTS AND LOCATIONS:
Overall Officials: Samir Y Saleh, PhD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Corvi F, Cozzi M, Barbolini E, Nizza D, Belotti M, Staurenghi G, Giani A. COMPARISON BETWEEN SEVERAL OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY DEVICES AND INDOCYANINE GREEN ANGIOGRAPHY OF CHOROIDAL NEOVASCULARIZATION. Retina. 2020 May;40(5):873-880. doi: 10.1097/IAE.0000000000002471. PMID 30807517
- [Result] Parravano M, Querques L, Scarinci F, Giorno P, De Geronimo D, Gattegna R, Varano M, Bandello F, Querques G. Optical coherence tomography angiography in treated type 2 neovascularization undergoing monthly anti-VEGF treatment. Acta Ophthalmol. 2017 Aug;95(5):e425-e426. doi: 10.1111/aos.13180. Epub 2016 Aug 6. No abstract available. PMID 27496070
- [Result] Grossniklaus HE, Green WR. Choroidal neovascularization. Am J Ophthalmol. 2004 Mar;137(3):496-503. doi: 10.1016/j.ajo.2003.09.042. PMID 15013874
- [Result] Querques G, Corvi F, Querques L, Souied EH, Bandello F. Optical Coherence Tomography Angiography of Choroidal Neovascularization Secondary to Pathologic Myopia. Dev Ophthalmol. 2016;56:101-6. doi: 10.1159/000442800. Epub 2016 Mar 15. PMID 27023343